CLINICAL TRIAL: NCT02609139
Title: A Phase 1, Open Label, Single-Dose, Within Cohort Randomized, 2-Way Crossover Study To Evaluate The Pharmacokinetics Of A Modified Release Formulation Of Pf-06650833 Under Fasting And Fed Conditions In Healthy Adult Subjects
Brief Title: Study to Evaluate Pharmacokinetics of A Modified Release Formulation of PF-06650833 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7921004; IRAK4 MR PK Study (Other: Alias Study Number)
Record Dates: First submitted 2015-11-05; First posted 2015-11-20 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- <=400mg Modified Release Tablets, Fasted (Experimental): Up to 400 mg PF-06650833 modified release tablets administered under fasted conditions
  Interventions: Drug: PF-06650833
- 100mg Modified Release Tablets, Fasted (Experimental): 100 mg PF-06650833 modified release tablets administered under fasted conditions
  Interventions: Drug: PF-06650833
- 20mg Modified Release Tablets, Fasted (Experimental): 20 mg PF-06650833 modified release tablets administered under fasted conditions
  Interventions: Drug: PF-06650833
- <= 400mg Modified Release Tablets, Fed (Experimental): Up to 400 mg PF-06650833 modified release tablets administered with high fat meal food intake
  Interventions: Drug: PF-06650833
- 100mg Modifed Release Tablets, Fed (Experimental): 100 mg PF-06650833 modified release tablets administered with high fat meal food intake
  Interventions: Drug: PF-06650833
- 20mg Modified Release Tablets, Fed (Experimental): 20 mg PF-06650833 modified release tablets administered with high fat meal food intake
  Interventions: Drug: PF-06650833

INTERVENTIONS:
Drug: PF-06650833 — Up to 400mg modified release tablets administered under fasted conditions
  Arms: <=400mg Modified Release Tablets, Fasted
Drug: PF-06650833 — 100mg modified release tablet administered under fasted conditions
  Arms: 100mg Modified Release Tablets, Fasted
Drug: PF-06650833 — 20mg modified release tablet administered under fasted conditions
  Arms: 20mg Modified Release Tablets, Fasted
Drug: PF-06650833 — Up to 400mg modified release tablets administered with high fat meal food intake
  Arms: <= 400mg Modified Release Tablets, Fed
Drug: PF-06650833 — 100mg modified released tablet administered with high fat meal food intake
  Arms: 100mg Modifed Release Tablets, Fed
Drug: PF-06650833 — 20 mg modified release tablet administered with high fat meal food intake
  Arms: 20mg Modified Release Tablets, Fed

SUMMARY:
This is a Phase 1, open-label, single-dose, within-cohort randomized, 2-way crossover study to evaluate the PK of orally administered PF-06650833 modified release tablets under fasted and high fat meal fed conditions in healthy subjects.

DETAILED DESCRIPTION:
This is the third study of PF-06650833. The goals of the study are to assess the PK in healthy subjects of single doses of modified release (MR) tablets of PF-06650833 when orally administered under fasting and high fat meal fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non childbearing potential and/or male subjects, between the ages of 18 and 55 years
2. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Personally signed and dated Informed Consent
4. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
2. Any condition possibly affecting drug absorption
3. Positive urine drug screen.
4. Heavy smokers
5. History of regular heavy alcohol consumption within 6 months of Screening.
6. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives
7. Screening supine blood pressure <=100 mm Hg (systolic) or<=50 mm Hg (diastolic) or>=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest.
8. Screening pulse (HR) >100 bpm after at least 5 minutes of rest.
9. Single supine 12 lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening.
10. Abnormal chest X ray
11. History of TB or active or latent or inadequately treated infection, positive Quantiferon TB test.
12. History of hepatitis or positive testing for human HIV,HepBsAg, HepBc Ab or HCVAb
13. Any medical history of disease [ie, Gilbert's disease] that has the potential to cause a rise in total bilirubin over the ULN
14. Clinical laboratory abnormalities including:

    * Creatine kinase >1.2 X ULN;
    * CK MB > ULN;
    * Serum myoglobin >1.2 X ULN;
    * Cardiac Troponin I (cTn I) > ULN of the laboratory reference range;
    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) >=2 x ULN, total serum bilirubin >=1.5 mg/dL;
    * Subjects with benign ethnic neutropenia;
    * Hemoglobin <=14 gm/dl (males) and <=13 gm/dL (females).
15. Nursing female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 28 days after the last dose of investigational product or longer based upon the compound's half life characteristics.
16. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product until discharge from the study at the end of Period 2.

    Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of investigational product. Acetaminophen/paracetamol should not be used. As an exception, ibuprofen may be used at doses of 200 to 400 mg orally every 6 hours as needed for up to 3 of 7 consecutive days.
17. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
18. History of sensitivity to heparin or heparin induced thrombocytopenia.
19. History of cancer (other than treated basal cell and squamous cell carcinoma of the skin) in the previous 5 years.
20. Previous exposure to PF 06650833.
21. Unwilling or unable to comply with the Lifestyle guidelines
22. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
23. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Maximum plasma concentration (Cmax) of PF-06650833
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration (AUClast) of PF-06650833
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Area under the plasma concentration versus time curve from time zero extrapolated to infinite time (AUCinf) of PF-06650833 (if data permit)
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Dose-normalized maximum plasma Cmax (Cmax(dn)) of PF-06650833
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Dose-normalized area under the plasma concentration versus time curve from time zero to the time of the last quantitfiable concentration (AUClast(dn)) of PF-06650833
Plasma pharmacokinetic parameters of PF-06650833 (if data permit) | Baseline to up to Day 14 (0 to +1) postdose
  Dose-normalized area under the plasma concentration versus time curve from time zero extrapolated to infinite time (AUCinf(dn)) of PF-06650833 (if data permit)

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Time post dose associated with the maximum plasma concentration (Tmax) of PF-06650833
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Terminal half life of PF-06650833 (if data permit)
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Lag time of plasma concentration of PF-06650833 (if data permit)
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Absorption rate constant of PF-06650833 (Ka) (if data permit)
Plasma pharmacokinetic parameters of PF-06650833 | Baseline to up to Day 14 (0 to +1) postdose
  Apparent Clearance (CL/F) of PF-06650833 (if data permit)
Plasma pharmacokinetic parameters of PF-06650833 | Baseline for up to Day 14 (0 to +1) postdose
  Apparent Volume of Distribution (Vz/F) of PF-06650833 (if data permit)
Treatment emergent adverse events and withdrawals | Baseline to up to Day 14 (0 to +1) postdose
  Incidence and severity of treatment emergent adverse events and withdrawals due to treatment emergent adverse events
Vital signs | Baseline to up to Day 14 (0 to +1) postdose
  Changes from baseline in vital signs (blood pressure, pulse rate, and respiratory rate)
Electrocardiogram parameters | Baseline to up to Day 14 (0 to +1) postdose
  Changes from baseline in electrocardiogram parameters (standard 12-lead ECG)
Clinical laboratory measurement | Baseline to up to Day 14 (0 to +1) postdose
  Changes from baseline in clinical laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7921004&StudyName=A%20Phase%201%2C%20Open%20Label%2C%20Single%E2%80%91dose%2C%20Within%20Cohort%20Randomized%2C%202%E2%80%91way%20Crossover%20Study%20To%20Evaluate%20The%20Pharmacokinetics%20Of%20A%20Modified%20Release%20Formulation%20Of%20Pf%E2%80%9106650833%20Under%20Fasting%20And%20Fed%20Conditions%20In%20Healthy%20Adult%20Subjects